CLINICAL TRIAL: NCT04165083
Title: KEYMAKER-U01 Substudy 2: A Phase 2, Umbrella Study With Rolling Arms of Investigational Agents in Combination With Pembrolizumab in Treatment Naïve Patients With PD-L1 Positive Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: KEYMAKER-U01 Substudy 2: Efficacy and Safety Study of Pembrolizumab (MK-3475) When Used With Investigational Agents in Treatment-naïve Participants With Anti-programmed Cell Death Receptor Ligand 1 (PD-L1) Positive Advanced Non-small Cell Lung Cancer (NSCLC) (MK-3475-01B/KEYMAKER-U01B)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-01B; MK-3475-01B (Other: MSD); KEYMAKER-U01B (Other: MSD); 2023-506933-32-00 (Registry Identifier: EU CT); U1111-1294-6518 (Registry Identifier: UTN); 2020-001627-14 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death Receptor 1 (PD-1, PD1); Programmed Cell Death Receptor Ligand 1 (PD-L1, PDL1); Programmed Cell Death Receptor Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + MK-4830 (Experimental): On Day 1 of each 3-week cycle, participants receive pembrolizumab 200 mg intravenously (IV) PLUS MK-4830 IV for a maximum of 35 cycles (approximately 2 years)
  Interventions: Biological: Pembrolizumab; Biological: MK-4830
- Pembrolizumab + MK-0482 (Experimental): On Day 1 of each 3-week cycle, participants receive pembrolizumab 200 mg intravenously (IV) PLUS MK-0482 IV for a maximum of 35 cycles (approximately 2 years)
  Interventions: Biological: Pembrolizumab; Biological: MK-0482

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
Biological: MK-4830 — IV infusion
  Arms: Pembrolizumab + MK-4830
Biological: MK-0482 — IV infusion
  Arms: Pembrolizumab + MK-0482

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab (MK-3475) in combination with MK-4830 in treatment-naïve participants with advanced squamous or non-squamous NSCLC that is PD-L1 positive.

This study is one of three pembrolizumab substudies being conducted under one pembrolizumab umbrella master protocol (MK-3475-U01/KEYMAKER-U01).

The pembrolizumab+ MK-0482 arm was added with Amendment 6.

DETAILED DESCRIPTION:
The master screening protocol is MK-3475-U01(KEYMAKER-U01) - NCT04165798

ELIGIBILITY:
Inclusion:

* Has a histologically- or cytologically-confirmed diagnosis of Stage IV squamous or non-squamous NSCLC
* Has non-squamous NSCLC and is not eligible for an approved targeted therapy
* Is able to provide archival tumor tissue sample collected either within 5 years or within the interval from completion of last treatment but before entering the screening period or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated obtained within 90 days of treatment initiation
* Has not received prior systemic treatment for metastatic NSCLC
* Has programmed cell death ligand 1 (PD-L1) tumor proportion score (TPS) ≥1%
* Is able to complete all screening procedures within the 35-day screening window.
* Male participants must agree to use contraception and refrain from donating sperm during the treatment period and for at least 120 days after the last dose of study treatment
* Female participants must not be pregnant or breastfeeding, and at least one of the following conditions apply:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to use contraception during the treatment period and for at least 120 days after the last dose of study treatment
* Has adequate organ function within 10 days of initiation of study treatment

Exclusion Criteria:

* Has a diagnosis of small cell lung cancer
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study treatment, or New York Heart Association Class III or IV congestive heart failure
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study
* Has had major surgery <3 weeks before the first dose of study treatment
* Has received prior radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study treatment
* Has received any prior immunotherapy and was discontinued from that treatment due to a severe or worse immune-related adverse event (irAE)
* Has had chemotherapy or biological cancer therapy within 4 weeks before the first dose of study treatment or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the AEs due to cancer therapeutics administered more than 4 weeks before the first dose of study treatment (including participants who had previous immunomodulatory therapy with residual irAEs)
* Has received a live vaccine within 30 days before the first dose of study treatment. Any licensed COVID-19 vaccine (including for Emergency Use) in a particular country is allowed as long as they are messenger ribonucleic acid (mRNA) vaccines, adenoviral vaccines, or inactivated vaccines. Investigational vaccines (ie, those not licensed or approved for Emergency Use) are not allowed
* Has received prior systemic cytotoxic chemotherapy or other targeted or biological antineoplastic therapy for metastatic disease.
* Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent or prior therapy targeting other immuno-regulatory receptors or mechanisms
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study treatment
* Has had a severe hypersensitivity reaction to treatment with monoclonal antibodies (including pembrolizumab) and/or any of their excipients
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  PFS is defined as the time from first dose of study treatment until either the earliest date of documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 27 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE) | Up to approximately 24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (39):
- United States (18):
  - Banner MD Anderson Cancer Center ( Site 0001), Gilbert, Arizona
  - City of Hope ( Site 0014), Duarte, California
  - UCSF Medical Center at Mission Bay ( Site 0007), San Francisco, California
  - Georgetown University ( Site 0036), Washington D.C., District of Columbia
  - University of Kentucky Markey Cancer Center ( Site 0019), Lexington, Kentucky
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 0003), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0002), Boston, Massachusetts
  - Oncology Hematology West, PC DBA Nebraska Cancer Specialists ( Site 0031), Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center ( Site 0016), Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0037), Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0034), New York, New York
  - Sanford Fargo Medical Center ( Site 0039), Fargo, North Dakota
  - Cleveland Clinic Main ( Site 0006), Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center ( Site 0015), Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania ( Site 0010), Philadelphia, Pennsylvania
  - Sanford Cancer Center ( Site 0038), Sioux Falls, South Dakota
  - The University of Texas MD Anderson Cancer Center ( Site 0009), Houston, Texas
- Hungary (3):
  - Petz Aladar Megyei Oktato Korhaz ( Site 0062), Győr, Győr-Moson-Sopron
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 0060), Budapest
- Israel (7):
  - Soroka Medical Center ( Site 0072), Beersheba
  - Rambam Health Care Campus-Oncology ( Site 0076), Haifa
  - Shaare Zedek Medical Center ( Site 0075), Jerusalem
  - Meir Medical Center ( Site 0071), Kfar Saba
  - Rabin Medical Center ( Site 0074), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0070), Ramat Gan
  - Sourasky Medical Center ( Site 0077), Tel Aviv
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi ( Site 0173), Florence, Firenze
  - IRCCS Ospedale San Raffaele ( Site 0171), Milan
  - Policlinico Gemelli di Roma ( Site 0174), Roma
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0152), Koszalin, West Pomeranian Voivodeship
- South Korea (3):
  - Seoul National University Bundang Hospital ( Site 0081), Seongnam-si, Kyonggi-do
  - Severance Hospital ( Site 0080), Seoul
  - Samsung Medical Center ( Site 0082), Seoul
- Spain (2):
  - ICO L Hospitalet ( Site 0090), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Quiron Madrid ( Site 0091), Madrid

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26227&tenant=MT_MSD_9011